CLINICAL TRIAL: NCT00111176
Title: Study of Thoracic Aortic Aneurysm Repair With the Zenith TX2 Endovascular Graft
Brief Title: STARZ-TX2 Clinical Study: Study of Thoracic Aortic Aneurysm Repair With the Zenith TX2 Endovascular Graft
Acronym: STARZ-TX2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Collaborators: William Cook Europe (Industry); William Cook Australia (Industry); MED Institute, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-536; 37010
Record Dates: First submitted 2005-05-17; First posted 2005-05-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Thoracic Aortic Aneurysm
Keywords: Thoracic Aortic Aneurysm; Descending; minimally invasive; endovascular; rupture; back pain; stent graft; endovascular aneurysm repair; aortic aneurysm; thoracic
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Rupture; Back Pain; Aortic Aneurysm | interventions — Endovascular Aneurysm Repair; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Endovascular Repair
  Interventions: Device: Endovascular repair
- 2 (Other): Surgical
  Interventions: Procedure: Surgical

INTERVENTIONS:
Device: Endovascular repair — Endovascular repair.
  Other Names: TEVAR
  Arms: 1
Procedure: Surgical — Surgical endovascular repair
  Arms: 2

SUMMARY:
The STARZ-TX2 trial (Study of Thoracic Aortic Aneurysm Repair with the Zenith TX2(R) TAA [Thoracic Aortic Aneurysm] Endovascular Graft) is a clinical trial approved by the United States Food and Drug Administration (FDA) to study the safety and effectiveness of the Zenith TX2 TAA Endovascular Graft in the treatment of thoracic aortic aneurysms / ulcers.

DETAILED DESCRIPTION:
The STARZ-TX2 trial (Study of Thoracic Aortic Aneurysm Repair with the Zenith TX2(R) TAA Endovascular Graft) is a clinical trial approved by the FDA to study the safety and effectiveness of the Zenith TX2(R) TAA Endovascular Graft in the treatment of thoracic aortic aneurysms / ulcers. Instead of making a large incision in the chest, the physician makes a small incision near the groin to insert and guide the graft into place in the aorta, relieving pressure on the aneurysm and helping to reduce the risk of rupture.

The Zenith TX2 TAA Endovascular Graft is a reinforced fabric tube that is sized to the length of the aorta that needs to be covered to seal off the aneurysm / ulcer. The graft is made of a polyester material like that used in open surgical repair. Standard surgical suture is used to sew the graft material to a frame of self-expanding stainless steel stents, which provide support. The materials used in the Zenith TX2 system have a long history of use in medical implants.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with aneurysms / ulcers of the descending thoracic aorta
* Patients who are candidates for either surgery or endovascular repair
* Patients at least 18 years old

Exclusion Criteria:

* Age < 18 years
* Patients with other medical condition (e.g., cancer, congestive heart failure) that may cause non-compliance with the protocol, confound the results, or with limited life expectancy (i.e., less than 2 years)
* Patients pregnant, breast-feeding, or planning on becoming pregnant within 24 months
* Patients unwilling or unable to comply with the follow-up schedule
* Patients unable or who refuse to give informed consent
* Patients simultaneously participating in another investigative device or drug study. (The patient must have completed the primary endpoint of any previous study at least 30 days prior to enrollment in this study.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2004-03; Primary Completion 2007-07 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The primary hypothesis for effectiveness is that patients treated with the Zenith TX2(R) TAA Endovascular Graft will have equivalent 30-day rupture-free survival compared to the surgical control. | 30 days

SECONDARY OUTCOMES:
A secondary hypothesis is subjects treated with the Zenith TX2(R) TAA Endovascular Graft will have equivalent or fewer complications compared to the surgical control group through 30 days following implant. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jon Matsumura, MD, Principal Investigator — University of Wisconsin, Madison
Locations (41):
- United States (38):
  - Banner Desert Medical Center, Mesa, Arizona
  - Arizona Heart Institute, Phoenix, Arizona
  - University of California, San Francisco, San Francisco, California
  - Stanford University Hospital and Clinics, Stanford, California
  - Swedish Medical Center, Englewood, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - St. Vincent Hospital, Indianapolis, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Union Memorial Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Albany Medical Center, Albany, New York
  - New York University Hospital, New York, New York
  - Lenox Hill Hospital, New York, New York
  - New York Presbyterian - Cornell, New York, New York
  - New York Presbyterian Hospital - Columbia, New York, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - MeritCare, Fargo, North Dakota
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- Canada (2):
  - Peter Lougheed Center, Calgary, Alberta
  - Vancouver Hospital and Health Science Center, Vancouver, British Columbia
- San Raffaele Hospital, Milan, Italy

REFERENCES:
- [Derived] Matsumura JS, Melissano G, Cambria RP, Dake MD, Mehta S, Svensson LG, Moore RD; Zenith TX2 Clinical Trial Investigators. Five-year results of thoracic endovascular aortic repair with the Zenith TX2. J Vasc Surg. 2014 Jul;60(1):1-10. doi: 10.1016/j.jvs.2014.01.043. Epub 2014 Mar 14. PMID 24636714